CLINICAL TRIAL: NCT01771731
Title: Cannabinoid-Based Therapy and Approaches to Quantify Pain in Sickle Cell Disease
Brief Title: Vaporized Cannabis for Chronic Pain Associated With Sickle Cell Disease
Acronym: Cannabis-SCD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: U54HL117664-01; 6610 (Other: UCSF Clinical and Translational Science Institute)
Record Dates: First submitted 2013-01-14; First posted 2013-01-18 (Estimated); Results first posted 2020-08-18 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — nabiximols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Cannabis (Experimental): Contents of 1 cannabis cigarette (4.7% THC/5.1% CBD) will be vaporized and inhaled at 12pm on Day 1; 8am, 2pm and 8pm on Days 2-4; and 8am on Day 5.
  Interventions: Drug: Cannabis
- Placebo (Placebo Comparator): Contents of 1 placebo cigarette (0% THC/0% CBD) will be vaporized and inhaled at 12pm on Day 1; 8am, 2pm and 8pm on Days 2-4; and 8am on Day 5.
  Interventions: Drug: Cannabis

INTERVENTIONS:
Drug: Cannabis
  Other Names: marijuana

SUMMARY:
Our primary objective is to assess whether inhaling vaporized cannabis ameliorates chronic pain in patients with sickle cell disease (SCD). As these patients will all be on chronic opioid analgesics, the investigators will also assess the possible synergistic affect between inhaled cannabis and opioids. The investigators will also assess the clinical safety of the concomitant use of cannabinoids and these opioids in patients with SCD by monitoring the short-term side effects associated with combined therapy. Finally, the investigators will evaluate the short-term effects of inhaled cannabis on markers of inflammation and disease progression in patients with SCD.

Hypotheses are as follows:

1. Inhaled cannabis will significantly reduce chronic pain in patients with SCD.
2. Inhaled cannabis will significantly alter the short-term side effects experienced by patients who take opioids for SCD.
3. Inhaled cannabis will significantly alter markers of inflammation and disease progression in patients with SCD compared to placebo.

DETAILED DESCRIPTION:
This is a proof-of-principle investigation of the safety and potential effectiveness of inhaled vaporized cannabis when added to a stable analgesic regimen in sickle cell disease (SCD) patients with chronic pain. The study will be comprised of two 5-day intervention periods in the inpatient setting (the Clinical Research Center at SFGH), with completion of a 5-day daily pain diary prior to admission to establish an outpatient baseline. Participants will be randomly assigned, in double-blind fashion, to treatment with (A) vaporized cannabis with an approximately 1:1 ration of delta-9-tetrahydrocannabinol:cannabidiol or (B) vaporized placebo. Those who receive treatment A during the first admission will receive treatment B in the second, and those who receive treatment B during the first admission will receive treatment A in the second. The two admissions will be spaced at least 14 days apart.

On Day 1 of each admission, subjects will provide blood samples for baseline markers of inflammation and SCD disease progression. They will undergo assessments of pain, mood, and quality of life. At 12 pm on Day 1, they will inhale vaporized study agent (equivalent to 1 cannabis/placebo cigarette) using the Volcano® vaporizer; on Days 2-4 they will inhale study agent at 8 am, 2 pm, and 8 pm, and they will inhale their final dose on Day 5 at 8 am. Subjects will continue their pre-study analgesic regimen while in the study. If additional analgesia is required, supplemental therapy will be administered and the dose recorded. Pain measurements by visual analogue scale will be obtained every 2 hours while subjects are awake. On Day 5 a second set of blood samples for inflammation markers and disease progression will be obtained, and subjects will again complete pain, mood, and quality of life assessments.

ELIGIBILITY:
Inclusion Criteria:

* Sickle cell disease, including sickle cell anemia (SS), sickle-hemoglobin C disease (SC), and sickle beta thalassemia disease (Sb).
* Ongoing opioid analgesic therapy for chronic sickle cell disease-associated pain.
* Subjects must be on a stable dose of analgesic medication (opioid or other) for at least 2 weeks before enrollment.
* All men and women in this study must agree to use adequate birth control during this study. Acceptable barrier birth control methods are a male condom, female condom, diaphragm, or intra-uterine (IUD).
* All women of reproductive potential (who have not reached menopause or undergone hysterectomy, oophorectomy, or tubal ligation) must have a negative urine b-HCG pregnancy test performed before initiating the protocol-specified medication.
* Prior history of use of cannabis. Subjects must have smoked cannabis on at least 6 occasions in their lifetime prior to enrollment.
* Subjects will self-report abstaining from smoking or ingesting cannabis for one week prior to their enrollment into the study.
* Able to understand and follow the instructions of the investigator, including completing the pain intensity rating scales.
* Karnofsky Performance Scale >60.
* Able and willing to provide informed consent.
* Able and willing to spend two separate periods of 5 days and 4 nights in the Clinical Research Center at SFGH.

Exclusion Criteria:

* Severe coronary artery disease, uncontrolled hypertension, cardiac ventricular conduction abnormalities, orthostatic mean blood pressure drop greater than 24 mmHg, severe chronic obstructive pulmonary disease.
* Evidence of clinically significant hepatic or renal dysfunction based on judgment of physician.
* Positive serum THC level on Day 1 of study.
* Active substance abuse (e.g., alcohol or injection drugs) as determined by urine toxicity screening.
* Neurologic dysfunction or psychiatric disorder severe enough to interfere with assessment of pain or sensory systems.
* Current use of smoked tobacco products.
* Women who are pregnant or breast-feeding may not take part in this study.
* Unable to read or speak English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-08; Primary Completion 2017-05-12 (Actual); Study Completion 2017-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald I Abrams, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States

REFERENCES:
- [Result] Abrams DI, Couey P, Dixit N, Sagi V, Hagar W, Vichinsky E, Kelly ME, Connett JE, Gupta K. Effect of Inhaled Cannabis for Pain in Adults With Sickle Cell Disease: A Randomized Clinical Trial. JAMA Netw Open. 2020 Jul 1;3(7):e2010874. doi: 10.1001/jamanetworkopen.2020.10874. PMID 32678452
- [Derived] Oniyangi O, Cohall DH. Phytomedicines (medicines derived from plants) for sickle cell disease. Cochrane Database Syst Rev. 2020 Sep 25;9(9):CD004448. doi: 10.1002/14651858.CD004448.pub7. PMID 32977351

RESULTS

PARTICIPANT FLOW:
Groups:
- Cannabis First, Then Placebo: This group received active THC:CBD cannabis during their first 5-day inpatient admission and placebo during the second admission.
- Placebo First, Then Cannabis: This group received placebo cannabis during their first 5-day inpatient admission and THC:CBD cannabis during the second.
Period: Overall Study
Arm/Group | Cannabis First, Then Placebo | Placebo First, Then Cannabis
Started | 13 | 14
Completed | 11 | 12
Not Completed | 2 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Adverse event: Pain Crisis | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Cannabis First, Then Placebo: Contents of 1 cannabis cigarette (4.7% THC/5.1% CBD) will be vaporized and inhaled at 12pm on Day 1; 8am, 2pm and 8pm on Days 2-4; and 8am on Day 5.
  Contents of 1 placebo cigarette (0% THC/0% CBD) will be vaporized and inhaled at 12pm on Day 1; 8am, 2pm and 8pm on Days 2-4; and 8am on Day 5.
- Placebo First, Then Cannabis: Contents of 1 placebo cigarette (0% THC/0% CBD) will be vaporized and inhaled at 12pm on Day 1; 8am, 2pm and 8pm on Days 2-4; and 8am on Day 5.
  Contents of 1 cannabis cigarette (4.7% THC/5.1% CBD) will be vaporized and inhaled at 12pm on Day 1; 8am, 2pm and 8pm on Days 2-4; and 8am on Day 5.
- Total: Total of all reporting groups
Arm/Group | Cannabis First, Then Placebo | Placebo First, Then Cannabis | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.7 (12.8) | 33.3 (8.7) | 36.4 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 6 | 5 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 11 | 24
  White | 0 | 0 | 0
  More than one race | 0 | 3 | 3
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Pain Rating Using Visual Analog Scale at Day 1 and Day 5
Description: Visual analog scale (VAS) used to assess pain. The scale range is 0-100, lower score means lower pain, higher score means higher pain.
Time Frame: Day 1 and Day 5
Population: All participants received both interventions.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Cannabis | Placebo
Number analyzed (Participants) | 23 | 23
score on a scale
  Day 1 | 40.5 [29.3 to 51.7] | 45.8 [34.3 to 57.3]
  Day 5 | 30.3 [19 to 41.6] | 38.5 [28.6 to 48.4]

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the two 5-day admission periods separated by one month
Arm/Group | Cannabis | Placebo
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 13/23 | 12/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cannabis (N=23) | Placebo (N=23)
Anxiety (Nervous system disorders) | 9 | 7
Sedation (Nervous system disorders) | 13 | 12
Disorientation (Nervous system disorders) | 2 | 3
Paranoia (Nervous system disorders) | 1 | 1
Confusion (Nervous system disorders) | 2 | 2
Dizziness (Nervous system disorders) | 6 | 3
Nausea (Nervous system disorders) | 4 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-09-07): https://cdn.clinicaltrials.gov/large-docs/31/NCT01771731/Prot_SAP_000.pdf